CLINICAL TRIAL: NCT04540354
Title: Personalised Risk scOre For Implantation of Defibrillators in Patients With Reduced LVEF≤35% and a Low Risk for Sudden Cardiac Death (PROFID-Reduced)
Brief Title: Personalised Risk scOre For Implantation of Defibrillators in Patients With Reduced LVEF≤35% and a Low Risk for Sudden Cardiac Death
Acronym: PROFID-Reduced
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design needs to be updated considering the lack of a risk predictor with acceptable predictive performance for the discrimination between high- and low-risk patients and the overall low sudden cardiac death risk as found in the data analysis
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LHI-2020-02; 847999 (Other Grant/Funding Number: European Union's Horizon 2020 research and innovation programme)
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Infarction; Heart Failure; Sudden Cardiac Death
Keywords: Myocardial Infarction; Heart Failure; Sudden Cardiac Death; Implantable Cardioverter Defibrillator; PROFID; Personalized Medicine
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The PROFID-Reduced trial is an open-label, blinded outcome assessment study. Thus, unblinding proce-dures for investigators are not applicable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Medical Therapy without ICD device therapy (Experimental): Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure and will not receive an ICD device
  Interventions: Drug: Optimal Medical Therapy (OMT)
- Optimal Medical Therapy with ICD device therapy (Active Comparator): Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure and will receive an ICD device
  Interventions: Drug: Optimal Medical Therapy (OMT); Device: Implantable cardioverter-defibrillator (ICD)

INTERVENTIONS:
Drug: Optimal Medical Therapy (OMT) — Patients will be treated according to Optimal Medical Therapy defined by the 2016 ESC guidelines for the management of acute and chronic heart failure.
Device: Implantable cardioverter-defibrillator (ICD) — An ICD consists of an electronic medical device and electrode leads. The surgery can be performed in local anaesthesia, but a short general anaesthesia is required if the ICD has to be tested giving the patient an electric shock. Besides the possibility to shock during arrhythmias the ICD can potentially terminate ventricular tachycardias by rapid pacing for short periods (small bursts of pacing).
  The subcutaneous defibrillator is an established and valid alternative to the conventional ICD for the preven-tion of SCD. According to current guidelines, the subcutaneous defibrillator should be considered as an alternative to transvenous defibrillators in patients with an indication for an ICD when pacing therapy for bradycardia support, cardiac resynchronisation or antitachycardia pacing is not needed.
  Arms: Optimal Medical Therapy with ICD device therapy

SUMMARY:
The objective of the study is to demonstrate that in post-MI patients with symptomatic heart failure who receive optimal medical therapy for this condition, and with reduced LVEF ≤ 35% but low risk for SCD according to a personalised risk score, optimal medical therapy without ICD implantation (index group) is not inferior to optimal medical therapy with ICD implantation (control group) with respect to all-cause mortality.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is a major public health problem, causing ~50% of cardiac fatalities and accounting for ~20% of all deaths in Europe. The majority of SCD cases are associated with coronary artery disease, mostly as a result of ventricular tachyarrhythmias (ventricular tachycardia and ventricular fibrillation) after previous myocardial infarction (MI). A predictor for increased risk of SCD after MI is a severely impaired heart function as expressed by a reduced left ventricular ejection fraction (LVEF). Based on this and on historical multi-national landmark trials, which found improved survival in patients with severely reduced LVEF who received an ICD, current clinical guidelines recommend prophylactic ICD implantation in post-MI patients with a LVEF ≤35% to improve overall survival by prevention of SCD.

Current practice of ICD implantation based solely on LVEF has significant limitations and results in substantial over- and undertreatment of patients. Furthermore, current clinical practice is substantially limited by the fact that it is based on out-dated evidence, a point already highlighted in the last version of the ESC guidelines for prevention of SCD. Indeed, since then, mortality and specifically SCD following MI has dramatically decreased. As a result, the risk for SCD has decreased significantly in the last decades rendering questionable whether the clinical benefits attributed to ICD implantation may not be much lower nowadays than that observed in the pivotal trials conducted 15-20 years ago. Due to the inherent risks and considerable costs of the ICD, detailed evaluation of the patient's risks and benefits of ICD implantation is required on a case-by-case basis - leading to a personalised rather than a "one-size-fits-all" treatment approach. To do so, identification of low-risk patients who would not benefit from ICD implantation in parallel with identification of post-MI patients who are at true high risk of SCD regardless of LVEF status is urgently needed. Thus, in sum-mary there is a compelling clinical need to identify patients at high individual risk for SCD in order to protect them effectively with ICD implantation but at the same time refrain from ICD implantation in patients with low individual risk for SCD.

The objective of the study is to demonstrate that in post-MI patients with symptomatic heart failure who receive optimal medical therapy for this condition, and with reduced LVEF ≤ 35% but low risk for SCD according to a personalised risk score, optimal medical therapy without ICD implantation (index group) is not inferior to optimal medical therapy with ICD implantation (control group) with respect to all-cause mortality.

PROFID-Reduced is a non-commercial, investigator-driven, prospective, parallel-group, randomised, open-label, blinded outcome assessment (PROBE), multi-centre, non-inferiority trial without dedicated investigational medical device (Proof of Strategy Trial) with two groups with 1:1 randomi-sation. It will be conducted in about 12 European countries with more than 150 clinical sites participating

The study is event driven and the number of randomised patients is estimated to be 2,480, required to collect 374 first primary outcome events within 30 months of mean follow-up.

Total study duration:

Enrolment of 30 months. All patients will be followed until 374 valid primary endpoints are reached (event-driven trial) which is expected about 15 months after last patient in. Total study duration of 47 months is expected which might be adapted based on a blinded interim analysis of the overall occurrence of the primary endpoint.

Individual study duration:

Expected median follow-up time will be about 30 months per patient with a minimum follow-up time of 15 months and a maximum follow-up time of presumably 45 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Documented history of myocardial infarction either as ST segment elevation myocardial infarction (STEMI) or as non-ST segment elevation myocardial infarction (NSTEMI).
* Symptomatic heart failure with NYHA class II or III.
* On Optimal Medical Therapy (OMT) for at least 3 months prior to enrolment.
* LVEF ≤ 35% at transthoracic echocardiography or cardiac magnetic resonance imaging (MRI).
* Predicted personalised annual risk of SCD according to the clinical risk calculator ≤2.5%.
* Signed informed consent.

Exclusion Criteria:

* Class I or IIa indication for implantation of an ICD for secondary prevention of sudden cardiac death and ventricular tachycardia (according to the 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death, see Appendix V).
* Ventricular tachycardia induced in an electrophysiologic study.
* Unexplained syncope when ventricular arrhythmia is suspected as the cause of syncope.
* Conclusive clinical indication for CRT (class I or IIa indication according to the 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure)
* Carrying any implanted cardiac pacemaker, defibrillator or CRT device.
* Violation of instruction for use (IFU) of the selected ICD device by at least one of the random group treatments.
* Hospitalised with unstable heart failure with NYHA class IV within 1 month prior to enrolment.
* Acute coronary syndrome or cardiac revascularization therapy by coronary angioplasty or coronary artery bypass grafting within 3 months prior to enrolment.
* Cardiac valve surgery or percutaneous cardiac valvular intervention such as transcatheter aortic valve replacement or transcatheter mitral valve repair performed within 3 months prior to enrolment.
* On the waiting list for heart transplantation.
* Any known disease that limits life expectancy to less than 1 year.
* Participation in another clinical trial, either within the 3 months prior to enrolment or still on-going (participation in sub-studies connected to this trial is permitted).
* Previous participation in PROFID-Reduced.
* Drug abuse or clinically manifest alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to the occurrence of all-cause death | Randomization to end of study (event-driven, expected about 15 months after last patient in)

SECONDARY OUTCOMES:
Time from randomisation to death from cardivascular causes | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Time from randomisation to sudden cardiac death | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Time from randomisation to first hospital readmissions for cardiovascular causes after randomisation | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Average length of stay in hospital during the study period | Randomization to end of study (event-driven, expected about 15 months after last patient in)
Quality of life (EQ-5D-5L) trajectories over time | At baseline and 6-month intervals thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Department of Electrophysiology, Leipzig Heart Center at University of Leipzig; Nikolaos Dagres, MD, Principal Investigator — Department of Electrophysiology, Leipzig Heart Center at University of Leipzig

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://profid-project.eu/